CLINICAL TRIAL: NCT05965570
Title: A Phase 1, Open-label, Fixed-sequence Study to Investigate the Effect of Clarithromycin, a Strong CYP3A4 Inhibitor, on Brensocatib Pharmacokinetics in Healthy Subjects
Brief Title: A Study to Investigate Effect of Clarithromycin, a Strong CYP3A4 Inhibitor, on Brensocatib Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS1007-109
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — brensocatib; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brensocatib + Clarithromycin (Experimental): Participants will receive a single oral dose of brensocatib in the morning on Days 1 and 13 after an overnight fast, and oral doses of clarithromycin, twice daily (BID), with food on Days 8 to 19. On Day 13, brensocatib will be coadministered with the morning dose of clarithromycin. Clarithromycin can be taken with food, with the exception of the morning dose on the day of coadministration with brensocatib (Day 13), which will be taken after an overnight fast.
  Interventions: Drug: Brensocatib; Drug: Clarithromycin

INTERVENTIONS:
Drug: Brensocatib — Oral tablets.
  Other Names: INS1007
Drug: Clarithromycin — Oral tablets.

SUMMARY:
The primary purpose of this study is to determine the effect of clarithromycin on the single-dose pharmacokinetics (PK) of brensocatib in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Females of nonchildbearing potential and males, of any race, between 18 and 65 years of age, inclusive, without current disease.
* Body mass index between 18.0 and 32.0 kilograms per square meter (kg/m^2), inclusive, and a total body weight ≥50 kilograms (kg).

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed; cholecystectomy will not be allowed).
* Positive serology test results for hepatitis B panel or hepatitis C antibody and/or reactive human immunodeficiency virus 1/2 test.
* Participants whose results are compatible with prior immunization for hepatitis B or natural immunity may be included at the discretion of the investigator.
* Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test at screening or check-in.
* Poor peripheral venous access. Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) of Brensocatib | Pre-dose and at multiple timepoints post-dose on Days 1 to 8, and Days 13 to 20
  The effect of clarithromycin on the single dose pharmacokinetics of brensocatib will be assessed in healthy participants.

SECONDARY OUTCOMES:
Number of Participants who Experienced at Least one Adverse Event (AE) | Up to Day 27
  Determination of the safety and tolerability of a single oral dose of brensocatib when administered alone and with clarithromycin in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No